CLINICAL TRIAL: NCT00637936
Title: Perioperative Oxygen Fraction - Effects on the PaO2/FiO2-Index During Laparotomy
Brief Title: Respiratory Effects of Perioperative Oxygen During General Anaesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Danish Medical Research Council (Other)
Responsible Party: Lars S Rasmussen, Dept.of Anaesthesia, Centre of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KF 02 306766-B
Record Dates: First submitted 2008-03-10; First posted 2008-03-18 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Laparotomy
Keywords: perioperative oxygen; respiratory complications
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Group 1 is given 30% oxygen during and 2 hours after surgery
  Interventions: Drug: Oxygen
- 2 (Active Comparator): Group 2 is given 80% during and 2 hours after surgery.
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Inspiratory fraction during anaesthesia

SUMMARY:
Aim: To investigate the effect of high intra- and postoperative oxygen concentration (80%, as opposed to normally 30%) on pulmonary gas exchange and other pulmonary complications after abdominal surgery.

Background: Previous studies have shown possible beneficial effects of high perioperative oxygen concentration on surgical wound infection and healing, but all pulmonary effects are not clarified. Change in perioperative PaO2/FiO2 and shunt-fraction, measured by a gas rebreathing technique, can describe pulmonary oxygenation. This could add knowledge to the pulmonary effects of high vs. normal oxygen concentration.

Primary hypothesis of study: Perioperative use of a 80% oxygen concentration reduces the PaO2/FiO2-index compared to 30% oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Laparatomy, elective

Exclusion Criteria:

* Inability to give informed consent
* Chemotherapy within 3 months
* Other surgery within 30 days(except surgery in local anaesthesia)
* Inability to keep oxygen saturation above 90% without supplemental oxygen (measured preoperatively by pulse oximetry)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change in PaO2/FiO2-index during general anaesthesia. | End of surgery.

SECONDARY OUTCOMES:
Change in PaO2/FiO2-index during general anaesthesia and postoperative recovery. | 1½ hour after surgery.
Atelectasis and Pneumonia | 14 days after surgery
Arterial oxygen saturation | 2 hours and 3 days after surgery.
Change in functional residual capacity (FRC) | 2 hours after surgery.
Change in effective pulmonary bloodflow | 2 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Meyhoff, MD, Study Director — Dept. of Anaesthesia, Centre of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark; Lars S Rasmussen, MD, PHD, DMSC, Study Chair — Dept. of Anaesthesia, Centre of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark; Steen Henneberg, MD,DMSC, Study Director — Dept.of Anaesthesia, The Juliane Marie Center, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark; Anne Kathrine Stæhr, Principal Investigator — Detp. of Anaesthesia, Centre of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark; Poul L Christensen, MD, Study Director — Dept. of Anaesthesia and Intensive Care, Copenhagen University Hospital, Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Staehr AK, Meyhoff CS, Henneberg SW, Christensen PL, Rasmussen LS. Influence of perioperative oxygen fraction on pulmonary function after abdominal surgery: a randomized controlled trial. BMC Res Notes. 2012 Jul 28;5:383. doi: 10.1186/1756-0500-5-383. PMID 22840231